CLINICAL TRIAL: NCT02193607
Title: Improved Reconstruction Pelvic Surgery With and Without Tension-free Vaginal Tape-obturator in Women With Occult Stress Urinary Incontinence(PTOS): a Randomized Controlled Trial
Brief Title: Outcomes of Pelvic Surgery With and Without Anti-incontinence Procedure in Occult Stress Urinary Incontinence Patients
Acronym: PTOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTOS-2014
Record Dates: First submitted 2014-06-19; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Pelvic Organ Prolapse; Stress Urinary Incontinence; Other Specified Urinary Incontinence
Keywords: Occult stress incontinence; Pelvic Organ Prolapse; Surgical Intervention; TVT-O(Tension-free vaginal tape-obturator); Improved Reconstructive Pelvic Surgery; Combined Surgery; Two-step Approach; Prophylactic Incontinence Procedure; Randomized Controlled Trial
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No TVT-O (Active Comparator): Improved reconstruction pelvic surgery
  Interventions: Procedure: Improved reconstruction pelvic surgery
- Combined surgery group (Experimental): Improved reconstruction pelvic surgery TVT-O procedure
  Interventions: Procedure: TVT-O; Procedure: Improved reconstruction pelvic surgery

INTERVENTIONS:
Procedure: TVT-O — Artificial mesh belt is placed in the middle urethra to provide support to remain no leak
  Arms: Combined surgery group
Procedure: Improved reconstruction pelvic surgery — Repair of severe pelvic organ prolapse with mesh.

SUMMARY:
1. To evaluate whether a standardized tension-free vaginal tape-obturator(TVT-O) procedure, when added to a planned improved reconstruction pelvic surgery, improves the rate of urinary stress continence in subjects with occult stress incontinence.
2. Observe the immediate and short-term complications, overall urinary tract function, and other aspects of pelvic health between subjects with and without a TVT-O procedure.

DETAILED DESCRIPTION:
The primary aim of this randomized study is evaluate whether a standardized TVT-O procedure, when added to a planned improved reconstruction pelvic surgery for the treatment of pelvic organ prolapse, improves the rate of urinary stress continence in subjects with occult stress incontinence. Secondary aims include comparison of immediate and short-term complications, overall urinary tract function, and other aspects of pelvic health between subjects with and without a TVT-O procedure. The value of preoperative urodynamic testing with prolapse reduction and 1 hour pad test will also be compared between subjects with and without a concomitant TVT-O procedure.

ELIGIBILITY:
Inclusion Criteria:

* In the absence of medical contraindications for improved pelvic floor reconstruction surgery and the TVT-O surgery
* Bulge of paries anterior vaginas stage III-IV
* Uterine prolapse stage II-II
* Without symptoms of stress urinary incontinence
* Screening tests of occult stress urinary incontinence(OSUI) should be positive
* ≥55 years old.

Exclusion Criteria:

* Pregnancy
* Illegible to follow up after surgery
* Previous surgery for stress urinary incontinence
* Unfinished data collection before surgery

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Stress incontinence | 3 months to 2 years post-operation
  Urine loss from physical activity such as coughing, sneezing or laughing.

SECONDARY OUTCOMES:
Immediate and short-term complications | Intraoperative and 2 years post-opeartion
  Immediate and short-term complications such as hemorrhage, bladder perforation and infection.
Overall urinary tract function | 3 months, 12 months and 2 years post-operation
  Overall urinary tract function: two validated questionnaires, standardized POP-Q measurements, urodynamic testing with prolapse reduction and 1 hour pad test.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Obstetrics and Gynecology Department, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wei JT, Nygaard I, Richter HE, Nager CW, Barber MD, Kenton K, Amundsen CL, Schaffer J, Meikle SF, Spino C; Pelvic Floor Disorders Network. A midurethral sling to reduce incontinence after vaginal prolapse repair. N Engl J Med. 2012 Jun 21;366(25):2358-67. doi: 10.1056/NEJMoa1111967. PMID 22716974
- [Background] Schierlitz L, Dwyer PL, Rosamilia A, De Souza A, Murray C, Thomas E, Hiscock R, Achtari C. Pelvic organ prolapse surgery with and without tension-free vaginal tape in women with occult or asymptomatic urodynamic stress incontinence: a randomised controlled trial. Int Urogynecol J. 2014 Jan;25(1):33-40. doi: 10.1007/s00192-013-2150-7. Epub 2013 Jun 28. PMID 23812579
- [Background] Brubaker L, Cundiff GW, Fine P, Nygaard I, Richter HE, Visco AG, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy with Burch colposuspension to reduce urinary stress incontinence. N Engl J Med. 2006 Apr 13;354(15):1557-66. doi: 10.1056/NEJMoa054208. PMID 16611949